CLINICAL TRIAL: NCT04771988
Title: Trans-arterial Radioembolization in Patients With Hepatocellular Carcinoma and Portal Vein Tumoral Thrombosis
Brief Title: Radioembolization for Hepatocellular Carcinoma With Portal Vein Tumoral Thrombosis
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Rita Golfieri, Chief of Radiology Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: Y90-2-LT-15-01
Record Dates: First submitted 2021-02-18; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; macrovascular invasion; portal vein thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: yttrium-90 radioembolization — selective/superselective treatment using resin microspheres labeled with Yttrium-90

SUMMARY:
In patients with hgepatocellular carcinoma (HCC) and portal vein tumoral thrombosis (PVTT), Sorafenib represents the treatment of choice but more recently, trans-arterial radioembolization (TARE) with yttrium-90 has been also proposed. A considerable percentage of such patients are not only able to achieve stability of the disease, but also to obtain a complete radiological response (CR). The possibility of achieving a CR might allow these patients to be listed for liver transplantation (LT), in order to cure not only the cancer but also the underlying cirrhosis that generated it.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of HCC;
2. age ≥ 18 years;
3. performance status according to Eastern Cooperative Oncology Group 0-1;
4. preserved liver function (Child-Pugh score ≤B7);
5. PVTT limited to the first order portal branch.

Exclusion Criteria:

1. any contraindication to TARE treatment;
2. macrovascular invasion extended to the main portal trunk and/or to the contralateral portal branch;
3. presence of extra-hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with HCC and PVTT presenting to our Institution
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-05-08 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Response to radioembolization | 6 months
  The primary endpoint of this study was to assess the effect of radioembolization in HCC patients with PVTT

SECONDARY OUTCOMES:
Overall survival | 5 years
  The secondary endpoint was overall survival (OS)
Progression-free survival | 5 years
  The secondary endpoint was progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: rita golfieri, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Bologna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lau WY, Sangro B, Chen PJ, Cheng SQ, Chow P, Lee RC, Leung T, Han KH, Poon RT. Treatment for hepatocellular carcinoma with portal vein tumor thrombosis: the emerging role for radioembolization using yttrium-90. Oncology. 2013;84(5):311-8. doi: 10.1159/000348325. Epub 2013 Apr 18. PMID 23615394
- [Result] Salem R, Lewandowski RJ, Mulcahy MF, Riaz A, Ryu RK, Ibrahim S, Atassi B, Baker T, Gates V, Miller FH, Sato KT, Wang E, Gupta R, Benson AB, Newman SB, Omary RA, Abecassis M, Kulik L. Radioembolization for hepatocellular carcinoma using Yttrium-90 microspheres: a comprehensive report of long-term outcomes. Gastroenterology. 2010 Jan;138(1):52-64. doi: 10.1053/j.gastro.2009.09.006. Epub 2009 Sep 18. PMID 19766639
- [Derived] Barros N, Ermel A, Mihaylov P, Lacerda M, Fridell J, Kubal C. Deceased Donor Liver Transplantation from a SARS-CoV-2-Positive Donor to a SARS-CoV-2-Positive Recipient. Liver Transpl. 2021 Dec;27(12):1849-1851. doi: 10.1002/lt.26253. Epub 2021 Sep 17. No abstract available. PMID 34351679